CLINICAL TRIAL: NCT02988661
Title: A Widespread Self-management Education Program to Reduce Health Disparities in African American Women With Systemic Lupus Erythematosus
Brief Title: Women Empowered to Live With Lupus Study
Acronym: WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cristina M Drenkard, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003656; R01MD010455 (NIH)
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Autoimmunity; Immune System Disorders
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Disease Self-management Program (CDSMP) (Active Comparator): A random sample of African American women with SLE selected from the Georgians Organized Against Lupus (GOAL) parent cohort will be used to recruit participants into the CDSMP. This group will be identified as the WELL Cohort.
  Interventions: Behavioral: Chronic Disease Self-management Program (CDSMP)
- Usual Care (No Intervention): African American women consented into the parent Georgians Organized Against Lupus (GOAL) cohort who have not been selected to be enrolled in the intervention will comprise the usual care group. This group will continue their longitudinal assessments as part or the GOAL cohort data collection efforts.

INTERVENTIONS:
Behavioral: Chronic Disease Self-management Program (CDSMP) — The CDSMP consists of 6 weekly classes of two and a half hours each one, for six weeks. A group of 10-16 people with different chronic conditions attend the classes together. Classes are facilitated by two certified leaders, one or both of whom are non-health professionals with chronic diseases. The workshop covers topics such as: 1) how to deal with frustration, fatigue, pain and isolation, 2) exercise for maintaining and improving strength, flexibility, and endurance, 3) communicating effectively with family, friends, and health professionals, 4) nutrition, 5) decision making, 6) appropriate use of medications and how to evaluate new treatments. Participants receive a companion book, Living a Healthy Life with Chronic Conditions, and an audio relaxation CD, Relaxation for Mind and Body.
  Other Names: Living Well with a Chronic Condition Workshop
  Arms: Chronic Disease Self-management Program (CDSMP)

SUMMARY:
The purpose of this research is to examine whether the Chronic Disease Self-management Program (CDSMP) would improve health outcomes and reduce health care use in African American women with systemic lupus erythematosus (SLE). The CDSMP is a generic, evidence-based self-management education program that has been shown to help people with chronic conditions to take control of their health problems. This study focuses on African American women with SLE because the CDSMP has not been widely studied in this population.

DETAILED DESCRIPTION:
The CDSMP is an evidence-based, community-based, generic self-management program that consists of 6 weekly classes of two and a half hours each one, for six weeks. CDSMP classes are facilitated by certified peer leaders. Because the CDSMP is widely disseminated and available to the adult U.S. population through community centers, it may be a suitable and accessible option for African Americans with SLE, even though it is not specifically tailored to SLE or to African Americans. As the CDSMP has been primarily evaluated in predominantly white middle-class seniors with more common diseases (e.g. osteoarthritis, diabetes), the effectiveness of the CDSMP in helping African American women to self-manage SLE is unknown.

This study will examine the effectiveness of the CDSMP to improve patient-reported outcomes and reduce health care utilization in African American women with lupus. Using a two-group longitudinal cohort design with participants sampled from a parent population-based SLE cohort in Georgia, investigators will examine behaviors, health and healthcare outcomes, and the extent to which individual characteristics modify the effectiveness of the CDSMP.

The Georgians Organized Against Lupus (GOAL), a longitudinal cohort of patients with a validated diagnosis of SLE, will be used to enroll participants into the intervention. A random sample of African American women with SLE selected from the parent GOAL cohort will be recruited into the WELL (Women Empowered to Live with Lupus) cohort. WELL participants will attend the CDSMP classes in the community, along with people with other chronic illnesses. WELL participants will be asked to attend the CDSMP in the community and answer questionnaires at 4 select time periods before and after the program. Investigators will follow participant's progress for up to 18 months after they attend the CDSMP.

African American women from the GOAL cohort non-selected to be assigned to the intervention will comprise the usual care group. Participants will continue their longitudinal assessments as part of the GOAL cohort data collection efforts. Changes in outcomes for up to 18 months will be compared between WELL participants and the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in the GOAL study

Exclusion Criteria:

* Participation in the Chronic Disease Self-Management Program (CDSMP) in the past five years
* Significant cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Drenkard, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Drenkard C, Easley K, Bao G, Dunlop-Thomas C, Lim SS, Brady T. Overcoming barriers to recruitment and retention of African-American women with SLE in behavioural interventions: lessons learnt from the WELL study. Lupus Sci Med. 2020 Jun;7(1):e000391. doi: 10.1136/lupus-2020-000391. PMID 32532797
- [Derived] Twumasi AA, Shao A, Dunlop-Thomas C, Drenkard C, Cooper HLF. Health service utilization among African American women living with systemic lupus erythematosus: perceived impacts of a self-management intervention. Arthritis Res Ther. 2019 Jun 25;21(1):155. doi: 10.1186/s13075-019-1942-7. PMID 31238992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Emory University in Atlanta, Georgia, USA. Participant enrollment began January 19, 2017 and the 18-month follow-up assessments were completed by February 26, 2021.
Groups:
- Chronic Disease Self-management Program (CDSMP): A random sample of African American women with systemic lupus erythematosus (SLE) selected from the Georgians Organized Against Lupus (GOAL) parent cohort was used to recruit participants into the chronic disease self-management program (CDSMP). This group is identified as the Women Empowered to Live with Lupus (WELL) Cohort.
- Usual Care: African American women consented into the parent Georgians Organized Against Lupus (GOAL) cohort who were not selected to be enrolled in the intervention will comprise the usual care group. This group will continue their longitudinal assessments as part or the GOAL cohort data collection efforts.
Period: Overall Study
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Started | 168 | 531
Completed | 165 | 447
Not Completed | 3 | 84
Not completed — Death | 2 | 18
Not completed — Lost to Follow-up | 0 | 33
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Unable to complete the 18-month survey | 1 | 27

BASELINE CHARACTERISTICS:
Groups:
- Chronic Disease Self-management Program (CDSMP): A random sample of African American women with SLE selected from the Georgians Organized Against Lupus (GOAL) parent cohort was used to recruit participants into the CDSMP. This group is identified as the WELL Cohort.
- Total: Total of all reporting groups
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care | Total
Number analyzed (Participants) | 168 | 531 | 699
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 151 | 473 | 624
  >=65 years | 17 | 58 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.3) | 47.3 (14.0) | 47.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 531 | 699
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 168 | 531 | 699
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 168 | 531 | 699
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 168 | 531 | 699

OUTCOME MEASURES:

1. Primary Outcome: Communication With Physician - Stanford 3Q Scale Score
Description: The Stanford 3Q Scale is a three-question measure that assesses communication between patients and physicians. The participant is asked to rank their responses using a 5-point Likert scale. Total scores range fro 0 to 5 and a higher score indicates better communication with physicians.
Time Frame: Baseline, Months 6, 12, and 18
Population: This analysis includes participants who completed the assessment at the indicated time points. Not all participants responded to all surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 522
score on a scale
  Baseline | 3.1 (1.1) | 2.9 (1.1)
  Month 6: number analyzed (Participants) | 156 | 263
  Month 6 | 3.3 (1.2) | 3.0 (1.1)
  Month 12: number analyzed (Participants) | 156 | 367
  Month 12 | 3.3 (1.1) | 3.0 (1.1)
  Month 18: number analyzed (Participants) | 165 | 442
  Month 18 | 3.3 (1.1) | 3.0 (1.1)

2. Primary Outcome: Patient-Reported Outcome Measurement Information System (PROMIS) Self-efficacy for Managing Medications and Treatments Score
Description: Self-efficacy for managing medical care was assessed with the PROMIS Self-efficacy for Managing Medications and Treatments Short Form (SF) 8a instrument. This is an eight-item tool that quantifies the level of current confidence (from 1=not confident at all to 5=very confident) a person with a chronic condition has in taking and managing medication and other treatments in challenging situations (e.g., traveling, running out of medication, occurrence of side effects). Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score indicates better self-efficacy for managing medications and treatments; scores higher than 50 indicate greater self-efficacy for managing medical care compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 524
T-score
  Baseline | 46.1 (9.1) | 46.1 (9.2)
  Month 6: number analyzed (Participants) | 156 | 265
  Month 6 | 47.0 (9.0) | 47.5 (8.5)
  Month 12: number analyzed (Participants) | 156 | 369
  Month 12 | 46.2 (8.8) | 47.0 (8.9)
  Month 18: number analyzed (Participants) | 165 | 447
  Month 18 | 45.9 (8.7) | 48.3 (9.2)

3. Primary Outcome: PROMIS Global Health Physical Health Domain Score
Description: The PROMIS for Global Health short form is a 10-item instrument representing multiple domains such as general health, quality of life, and mental health. Participants will be asked to respond to questions on a scale from 1 to 5, where 1 represents poor health, and 5 represents excellent health. Total raw scores are calculated for two domains: Physical Health and Mental Health. Raw scores are further converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates better physical health; scores higher than 50 indicate greater physical health compared to the reference population..
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 166 | 530
T-score
  Baseline | 38.3 (7.5) | 40.6 (8.8)
  Month 6: number analyzed (Participants) | 153 | 265
  Month 6 | 39.0 (7.5) | 40.0 (8.6)
  Month 12: number analyzed (Participants) | 150 | 370
  Month 12 | 38.9 (7.6) | 40.3 (8.7)
  Month 18: number analyzed (Participants) | 160 | 446
  Month 18 | 39.1 (7.5) | 40.3 (8.8)

4. Primary Outcome: PROMIS Global Health Mental Health Domain Score
Description: The PROMIS for Global Health short form is a 10-item instrument representing multiple domains such as general health, quality of life, and mental health. Participants will be asked to respond to questions on a scale from 1 to 5, where 1 represents poor health, and 5 represents excellent health. Total raw scores are calculated for two domains: Physical Health and Mental Health. Raw scores are further converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates better mental health; scores higher than 50 indicate better mental health compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 166 | 530
T-score
  Baseline | 41.5 (8.9) | 43.5 (9.3)
  Month 6: number analyzed (Participants) | 153 | 265
  Month 6 | 42.4 (9.1) | 43.2 (8.8)
  Month 12: number analyzed (Participants) | 150 | 370
  Month 12 | 42.4 (8.6) | 43.4 (9.1)
  Month 18: number analyzed (Participants) | 160 | 446
  Month 18 | 42.3 (7.9) | 43.6 (9.3)

5. Primary Outcome: PROMIS Physical Function Score
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function SF 10b is a self-administered instrument that assesses self-reported capability rather than actual performance of physical activities. Participants are asked to respond to questions regarding the extent of their physical function. Responses range from 1 to 5, where 1 represents "unable to do" and 5 represents "without any difficulty". Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates better physical function capabilities; scores higher than 50 indicate greater physical function compared to the reference population.
Time Frame: Baseline, Months 6, 12, 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 528
T-score
  Baseline | 38.4 (7.6) | 40.5 (10.0)
  Month 6: number analyzed (Participants) | 155 | 267
  Month 6 | 38.4 (7.6) | 40.8 (9.8)
  Month 12: number analyzed (Participants) | 155 | 370
  Month 12 | 39.0 (8.4) | 40.1 (9.9)
  Month 18: number analyzed (Participants) | 164 | 447
  Month 18 | 38.4 (7.5) | 40.4 (9.8)

6. Primary Outcome: PROMIS Pain Interference Score
Description: The PROMIS Pain Interference SF 8a is a self-administered instrument that assesses the interference of pain on daily activities. Participants are asked to respond to questions regarding the extent of their pain. Responses range from 1 to 5, where 1 represents "not at all" and 5 represents "very much". Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A lower score indicates the least amount of pain interference; scores higher than 50 indicate greater pain interference compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 167 | 527
T-score
  Baseline | 59.0 (9.2) | 57.7 (10.1)
  Month 6: number analyzed (Participants) | 155 | 267
  Month 6 | 59.1 (9.0) | 57.6 (10.0)
  Month 12: number analyzed (Participants) | 156 | 370
  Month 12 | 59.3 (8.7) | 57.9 (10.7)
  Month 18: number analyzed (Participants) | 165 | 446
  Month 18 | 59.3 (8.6) | 58.1 (10.1)

7. Primary Outcome: PROMIS Fatigue Score
Description: The PROMIS Fatigue SF 8a is a self-administered instrument that assesses fatigue level within the past seven days. Participants are asked to respond to questions regarding fatigue frequency. Responses range from 1 to 5, where 1 represents "never" and five represents "always". Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10; scores higher than 50 indicate greater fatigue compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 523
T-score
  Baseline | 58.6 (10.5) | 57.6 (11.2)
  Month 6: number analyzed (Participants) | 156 | 266
  Month 6 | 59.5 (9.7) | 57.5 (11.3)
  Month 12: number analyzed (Participants) | 155 | 369
  Month 12 | 58.7 (10.0) | 57.8 (11.0)
  Month 18: number analyzed (Participants) | 164 | 446
  Month 18 | 58.2 (10.5) | 57.4 (11.3)

8. Primary Outcome: PROMIS Sleep Disturbance Score
Description: The PROMIS Sleep Disturbance SF 8a is a self-administered instrument to assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. It assesses sleep disturbance over the past seven days. Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates more sleep disturbance; scores higher than 50 indicate greater sleep disturbance compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 526
T-score
  Baseline | 57.3 (10.8) | 56.6 (10.8)
  Month 6: number analyzed (Participants) | 156 | 267
  Month 6 | 57.8 (10.0) | 55.8 (10.1)
  Month 12: number analyzed (Participants) | 155 | 370
  Month 12 | 57.3 (10.3) | 56.5 (10.1)
  Month 18: number analyzed (Participants) | 165 | 447
  Month 18 | 57.7 (9.8) | 55.0 (9.0)

9. Primary Outcome: PROMIS Anxiety Score
Description: The PROMIS Anxiety SF 8a is a self-administered instrument to assess emotional distress within the past seven days. Participants are asked to rate their anxiety level for various items ranked from 1 to 5, where 1 represents "never" and 5 represents "always". Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates high anxiety; scores higher than 50 indicate greater anxiety compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 526
T-score
  Baseline | 53.8 (10.5) | 52.0 (11.5)
  Month 6: number analyzed (Participants) | 156 | 267
  Month 6 | 54.6 (10.4) | 50.5 (11.1)
  Month 12: number analyzed (Participants) | 156 | 370
  Month 12 | 54.3 (10.6) | 52.0 (11.2)
  Month 18: number analyzed (Participants) | 163 | 445
  Month 18 | 53.2 (10.7) | 51.6 (11.3)

10. Primary Outcome: PROMIS Ability to Participate in Social Roles and Activities Score
Description: The PROMIS Ability to Participate in Social Roles and Activities SF 8a is a self-administered instrument to assess perceived ability to perform one's usual social roles and activities. Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates better perceived abilities; scores higher than 50 indicate better perceived abilities to participate in social activities and roles compared to the reference population.
Time Frame: Baseline, Months 6, 12, 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 520
T-score
  Baseline | 45.3 (8.3) | 47.4 (10.1)
  Month 6: number analyzed (Participants) | 156 | 267
  Month 6 | 45.0 (8.7) | 47.1 (10.2)
  Month 12: number analyzed (Participants) | 155 | 370
  Month 12 | 45.5 (8.5) | 46.6 (10.0)
  Month 18: number analyzed (Participants) | 164 | 447
  Month 18 | 45.5 (8.1) | 47.0 (9.6)

11. Secondary Outcome: Number of Participants at Each Activation Level of the Patient Activation Measure (PAM-10)
Description: The Patient Activation Measure (PAM-10) is a 10-item tool to assess an individual's knowledge, skill, and confidence for managing one's health and healthcare. Individuals who measure high on this assessment typically understand the importance of taking a pro-active role in managing their health and have the skills and confidence to do so. The PAM-10 survey measures individuals activation on a 0-100 scale, which are further grouped in 4 levels of activation along an empirically derived continuum. Activation Level 1 is "Disengaged & Overwhelmed" where knowledge of and adherence to healthcare and is low. Activation Level 2 is "Becoming Aware But Still Struggling" where individuals can set simple goals but believe health is out of their control. Activation Level 3 is "Taking Action & Gaining Control" where individuals are building self-management skills. Activation Level 4 is "Maintaining Behaviors & Pushing Further" where individuals are maintaining newly adopted behaviors.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 165 | 523
Participants
  Baseline: Level 1: Disengaged & Overwhelmed | 12 | 40
  Baseline: Level 2: Becoming Aware But Still Struggling | 25 | 123
  Baseline: Level 3: Taking Action & Gaining Control | 72 | 206
  Baseline: Level 4: Maintaining Behaviors & Pushing Further | 56 | 154
  Month 6: number analyzed (Participants) | 154 | 260
  Month 6: Level 1: Disengaged & Overwhelmed | 13 | 25
  Month 6: Level 2: Becoming Aware But Still Struggling | 26 | 44
  Month 6: Level 3: Taking Action & Gaining Control | 56 | 101
  Month 6: Level 4: Maintaining Behaviors & Pushing Further | 59 | 90
  Month 12: number analyzed (Participants) | 154 | 366
  Month 12: Level 1: Disengaged & Overwhelmed | 8 | 26
  Month 12: Level 2: Becoming Aware But Still Struggling | 13 | 73
  Month 12: Level 3: Taking Action & Gaining Control | 70 | 154
  Month 12: Level 4: Maintaining Behaviors & Pushing Further | 63 | 113
  Month 18: number analyzed (Participants) | 164 | 436
  Month 18: Level 1: Disengaged & Overwhelmed | 14 | 33
  Month 18: Level 2: Becoming Aware But Still Struggling | 30 | 80
  Month 18: Level 3: Taking Action & Gaining Control | 58 | 161
  Month 18: Level 4: Maintaining Behaviors & Pushing Further | 62 | 162

12. Secondary Outcome: PROMIS Adult Self-Efficacy Score
Description: The PROMIS Adult Self-Efficacy SF 4a is a self-administered instrument to assess current level of confidence in managing symptoms of chronic conditions. Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates higher self-efficacy; scores higher than 50 indicate greater self-efficacy compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 522
T-score
  Baseline | 47.1 (7.8) | 48.4 (8.7)
  Month 6: number analyzed (Participants) | 156 | 264
  Month 6 | 47.5 (7.8) | 49.1 (9.0)
  Month 12: number analyzed (Participants) | 156 | 366
  Month 12 | 48.2 (8.5) | 48.7 (8.6)
  Month 18: number analyzed (Participants) | 165 | 446
  Month 18 | 48.2 (7.8) | 49.3 (8.8)

13. Secondary Outcome: PROMIS Anger Score
Description: The PROMIS Anger SF 5a is a self-administered instrument to measure angry mood (irritability, frustration), negative social cognitions (interpersonal sensitivity, envy, disagreeableness), and efforts to control anger. Total raw scores are converted to T-scores by the Health Measures Scoring Service. The T-score rescales the raw score into a standardized score with a mean of 50 and an SD of 10. A higher score indicates more anger; scores higher than 50 indicate greater anger compared to the reference population.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 522
T-score
  Baseline | 53.2 (11.6) | 51.0 (12.4)
  Month 6: number analyzed (Participants) | 156 | 267
  Month 6 | 53.5 (13.0) | 50.3 (12.5)
  Month 12: number analyzed (Participants) | 156 | 370
  Month 12 | 52.7 (11.8) | 50.8 (12.3)
  Month 18: number analyzed (Participants) | 165 | 445
  Month 18 | 52.3 (12.3) | 50.9 (12.6)

14. Secondary Outcome: Perceived Stress Scale 4 (PSS-4) Score
Description: The Perceived Stress Scale 4 (PSS-4) is the most widely used psychological instrument for measuring the perception of stress. Participants are asked to rank responses to each of the four items on a scale from 0 to 4, where zero means never and four means very often. Total scores range from 0 to 16 and a higher score indicates higher perceived stress.
Time Frame: Baseline, Months 6, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 526
score on a scale
  Baseline | 6.2 (3.2) | 6.3 (3.2)
  Month 6: number analyzed (Participants) | 156 | 267
  Month 6 | 6.2 (3.3) | 6.1 (3.2)
  Month 12: number analyzed (Participants) | 156 | 368
  Month 12 | 6.0 (3.3) | 6.4 (3.1)
  Month 18: number analyzed (Participants) | 165 | 446
  Month 18 | 6.1 (3.2) | 6.1 (3.1)

15. Secondary Outcome: Hospitalization Rate
Description: The number of hospitalizations were collected from the Georgia Department of Public Health (DPH) administrative data for the pre- and post-intervention period (up to two years). The hospitalization rate is the hospitalizations per 100 person years, adjusted for mortality and leaving the state of Georgia. For participants in the CDSMP group, data were collected for the period of one year before and one year after the date when the CDSMP workshop started. For participants receiving usual care, data were collected one year before and one year after the index date, which is when 50% of CDSMP participants started their first intervention class.
Time Frame: One year before and one year after the start of the study intervention (up to 2 years)
Population: This analysis includes participants with data available with the Georgia Department of Public Health.
Measure: Number; unit: hospitalizations per 100 person years
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 531
hospitalizations per 100 person years
  During the year before the start of the study intervention: number analyzed (Participants) | 168 | 516
  During the year before the start of the study intervention | 42.3 | 45.5
  During the year after the start of the study intervention | 49.6 | 47.8

16. Secondary Outcome: Emergency Department Visit Rate
Description: The number of emergency department (ED) visits were collected from the Georgia DPH administrative data for the pre- and post-intervention period (up to two years). The emergency department visit rate is the emergency department visits per 100 person years, adjusted for mortality and leaving the state of Georgia. For participants in the CDSMP group, data were collected for the period of one year before and one year after the date when the CDSMP workshop started. For participants receiving usual care, data were collected one year before and one year after the index date, which is when 50% of CDSMP participants started their first intervention class.
Time Frame: One year before and one year after the start of the study intervention (up to 2 years)
Population: This analysis includes participants with data available with the Georgia Department of Public Health.
Measure: Number; unit: ED visits per 100 person years
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
Number analyzed (Participants) | 168 | 531
ED visits per 100 person years
  During the year before the start of the study intervention: number analyzed (Participants) | 168 | 516
  During the year before the start of the study intervention | 126.2 | 121.3
  During the year after the start of the study intervention | 103.9 | 111.5

ADVERSE EVENTS:
Time Frame: Information concerning mortality was collected beginning at the baseline assessment and continued through the 18-month assessment.
Description: The intervention is a well-established education self-management program, consequently, adverse events were not expected to occur from participating in the study and were not collected. Nevertheless, information on all-cause mortality was collected beginning at the baseline assessment and continued through the 18-month assessment.
Arm/Group | Chronic Disease Self-management Program (CDSMP) | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/168 | 18/531
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT02988661/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02988661/ICF_001.pdf